CLINICAL TRIAL: NCT01908634
Title: A Pilot Study to Test the Effects of Matrix on Fruit Constituent Bioavailability and Influence on Chronic Disease Risk Factors.
Brief Title: Matrix on Fruit Constituent Bioavailability
Acronym: FRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 2013-076
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Results first posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Healthy Non-smoker
Keywords: Bioavailability; Strawberry polyphenols; Fruit Beverage Matrix
MeSH Terms: interventions — Meals

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Milk-based Strawberry Beverage no meal (Active Comparator): Milk-based Strawberry beverage without meal
  Interventions: Dietary Supplement: Milk-based Strawberry Beverage without meal
- Water-based Strawberry Beverage no meal (Experimental): Water-based Strawberry beverage without meal
  Interventions: Dietary Supplement: Water-Based Strawberry Beverage without meal
- Milk-based strawberry Beverage with meal (Active Comparator): Milk-based Strawberry beverage with meal
  Interventions: Dietary Supplement: Milk-based strawberry Beverage with meal
- Water-based strawberry Beverage with meal (Experimental): Water-based Strawberry beverage with meal
  Interventions: Dietary Supplement: Water-Based strawberry Beverage with meal

INTERVENTIONS:
Dietary Supplement: Milk-based Strawberry Beverage without meal
  Arms: Milk-based Strawberry Beverage no meal
Dietary Supplement: Water-Based Strawberry Beverage without meal
  Arms: Water-based Strawberry Beverage no meal
Dietary Supplement: Milk-based strawberry Beverage with meal
  Arms: Milk-based strawberry Beverage with meal
Dietary Supplement: Water-Based strawberry Beverage with meal
  Arms: Water-based strawberry Beverage with meal

SUMMARY:
Primary objective is to evaluate the influence of matrix on the bioavailability of key phytochemical constituents in fruits and their subsequent effect on chronic disease risk factors.

DETAILED DESCRIPTION:
This study is a single-center, randomized, cross-over, 4-arm, single- blinded, 6-hour postprandial study to evaluate the effects of strawberry or comparator fruit provided in a formulated beverage with milk (as the base) or water or fresh/pureed.

A planned sample size of 10 men and women will be recruited into the study. Subjects will be required to meet several inclusion and exclusion criteria, which will be assessed through online and clinic screening mechanisms, including questionnaires, fasting glucose concentration, and anthropometric measurements. Eligible subjects will be invited to participate in the study. Subjects will begin by completing a 3-day pre-study assessment of their usual dietary intake using 3-day food diary. After reviewing baseline food records, subjects will be instructed to avoid polyphenolic-containing foods for 2 days prior to the study visit, while maintaining their usual diet pattern and physical activity.

Subjects will participate in 6 h postprandial study days. Subjects will be randomized on the first day of starting the first post prandial visit day.

For each 6 h postprandial study visit, subjects will arrive fasted and follow procedures published by our lab previously. This includes: pre-study evaluation for compliance (fasting, dinner consumption, limited polyphenol intake) and readiness for study visit, catheter placement by registered nurse, fasting blood sample, consumption of high fat/carbohydrate meal accompanied by 1 of the treatment beverages, subsequent blood sampling from catheter [ ~1 tablespoon (12ml)] at designated time points for 6 hours.

Each postprandial study visit day will last approximately 7 hours and subjects will be required to remain at the Clinical Nutrition Research Center at the Illinois Institute of Technology main campus for the duration of the visit. The visit procedures are repeated four times ~ 1 week apart to accommodate subject testing with all four beverages; all procedures are identical on each postprandial study test visit with the exception that only an assigned test beverage per each visit will be consumed with the breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-78 years of age)
* Relatively healthy
* Non-smoker or past smoker with abstinence for at least 2 years

Exclusion Criteria:

* Pregnant and/or breast feeding
* Smoker or past smoker with abstinence <2 years
* Allergy or intolerance to study foods
* Current regular consumption of berries is > 2 servings per day.
* Fasting blood glucose ≥ 126 mg/dL. Subjects identified with elevated fasting blood glucose levels will be advised to contact their primary care physician for appropriate follow-up care.
* Taking over the counter antioxidant supplements or other supplements that may interfere with the study procedures or endpoints.
* Subjects with unusual dietary habits (e.g. pica).
* Actively losing weight or trying to lose weight (unstable body weight fluctuations of > 5 lbs in a 60 day period).
* Excessive exercisers or trained athletes.
* Subjects with documented atherosclerotic disease, inflammatory disease, diabetes mellitus, or other systemic diseases.
* Addicted to drugs and/or alcohol.
* Medically documented psychiatric or neurological disturbances.
* Severe obesity as defined by >39.9 BMI or under weight for height (BMI <18.5)

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Relatively healthy individuals were screened and recruited in Chicago, IL for the study at the Clinical Nutrition Research Center (CNRC) from 2013 to 2014
Pre-assignment Details: Eligible participants followed a low polyphenol diet 3 days before each test day visit (3 days run-in), while maintaining their usual diet and physical activity patterns.
Groups:
- All Participants: All participants received multiple interventions in *1* sequence (i.e., Water-based Strawberry Beverage With Meal first, then Milk-based Strawberry Beverage With Meal, then Water-based Strawberry Beverage Without Meal, then Milk-based Strawberry Beverage Without Meal)
Period: Milk-based Strawberry Beverage With Meal
Arm/Group | All Participants
Started | 10
Completed (cross over design) | 10
Not Completed | 0
Period: Water-based Strawberry Beverage Wit Meal
Arm/Group | All Participants
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Milk-based Strawberry Beverage w/o Meal
Arm/Group | All Participants
Started | 9
Completed | 4
Not Completed | 5
Not completed — Withdrawal by Subject | 5
Period: Water-based Strawberry Beverage w/o Meal
Arm/Group | All Participants
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants, measured at screening visit
Arm/Group | All Participants
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years]
  All | 24.5 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: CMax in Polyphenol Anthocyanin Concentrations
Description: Changes in Plasma polyphenol anthocyanin concentrations over 6 hr (from 0 to 6 hrs), assessed by time and treatment effect Cmax
Time Frame: 6 hours
Population: Nine subjects completed Part 1 (beverage with meal) and a subset of 4 completed Part 2 (beverages without meal).
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Milk-based Strawberry Beverage no Meal | Water-based Strawberry Beverage no Meal | Milk-based Strawberry Beverage With Meal | Water-based Strawberry Beverage With Meal
Number analyzed (Participants) | 4 | 4 | 9 | 9
nmol/L | 8.7 (0.7) | 22.1 (3.8) | 7.6 (1.5) | 11.3 (2.7)

ADVERSE EVENTS:
Time Frame: up to 6 weeks
Groups:
- Without Meal: Milk-based strawberry Beverage without a meal vs. Water-based strawberry Beverage without a meal
- With Meal: Milk-based strawberry Beverage with a meal vs. Water-based strawberry Beverage with a meal
Arm/Group | Without Meal | With Meal
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/9
Other Adverse Events (participants affected / at risk) | 0/4 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No